CLINICAL TRIAL: NCT00253175
Title: A Comparison Of The Efficacy And Safety Of Topamax® (Topiramate) Tablets Versus Placebo For The Prophylaxis Of Migraine
Brief Title: A Study of the Effectiveness and Safety of Topiramate for the Prevention of Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005572
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Vascular Headaches; Migraine
Keywords: topiramate; migraine headache; migraine prevention; migraine
MeSH Terms: conditions — Vascular Headaches; Migraine Disorders | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness and safety of topiramate (an epilepsy medication) compared with placebo in the prevention of migraine.

DETAILED DESCRIPTION:
Topiramate is a medication that is widely used for the treatment of adult and pediatric patients with seizures and has been shown in preliminary studies to be effective for migraine prevention in adults. This is an outpatient, randomized, double-blind, placebo-controlled study to confirm preliminary studies of the effectiveness of topiramate in the prevention of migraine attacks. The study is composed of 4 phases: pretreatment, double-blind treatment for 20 weeks, a blinded transition, and an open-label extension. During the pretreatment phase patients discontinue all medication for migraine prevention and keep a daily record of headache information in a diary. Patients with 3 to 8 migraines, but not more than 15 headache days, during the pretreatment phase continue in the double-blind treatment phase. In the 20-week double-blind treatment phase, oral topiramate tablets (or placebo) are taken daily beginning at 25 mg once daily for 1 week, increasing to twice daily doses of up to a maximum of 8 tablets (200 mg) per day during the 8-week titration period, and maintained at that dose during the 12-week maintenance period. Patients who successfully complete the double-blind therapy phase may continue in an open-label extension (32 weeks), during which the study medication (topiramate or placebo) will be decreased and simultaneously topiramate (open-label) will be administered at increasing doses. During the study, patients will maintain headache and medication records to document the following: occurrence and duration of headaches; severity of headache pain; associated symptoms, such as nausea, vomiting, photophobia (avoidance and dread of light), phonophobia (fear of sound); and medication taken to relieve headache pain or symptoms. The primary measure of effectiveness is the percent reduction in the frequency of monthly migraine episodes during the entire double-blind treatment phase compared with the pretreatment phase. Other assessments of effectiveness include the percent of patients responding to treatment (>= 50% reduction in average monthly migraine attacks) during the double-blind treatment phase compared with the pretreatment phase, the reduction in number of migraine days/month during treatment, and the reduction in severity and duration of migraines during treatment. Safety assessments include the incidence of adverse events throughout the study, and measurement of vital signs (pulse, blood pressure, body weight), physical examinations, and clinical laboratory tests (hematology, biochemistry, and urinalysis) at specified intervals. The study hypothesis is that the decrease in the mean monthly migraine rate is greater in the topiramate group than in the placebo group.

Oral topiramate tablets 25 mg or placebo tablets, beginning at 25 mg once daily for 1 week, increasing to twice daily doses of up to a maximum of 8 tablets (200 mg) during the 8-week titration period, and maintained at that dose during the 12-week maintenance period (20 weeks total duration).

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria of the International Headache Society for the classification of migraine with or without aura (migraine symptoms)
* Diagnosis of migraine for at least 12 months prior to start of the study
* Have had an average of 3 to 8 migraine attacks per month for the 3 months prior to the start of the study
* Ability to recognize migraine headaches and to distinguish them from tension-type headaches or other types of head pain
* General good health

Exclusion Criteria:

* Patients who previously failed to respond to topiramate therapy for migraine prevention or who discontinued topiramate due to adverse events
* Patients who had onset of migraine after age 50
* Patients having more than 15 headache-days per month during the 3 months prior to start of the study, or during the baseline (pretreatment) period
* Patients who have cluster headaches or who have exclusively aura (migraine symptoms) without headache
* Female patients who are pregnant, nursing, or those not using adequate birth control, if capable of bearing children

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2000-10; Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Reduction in the frequency of monthly migraine episodes during the entire double-blind treatment phase compared with the pretreatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Silberstein SD, Hulihan J, Karim MR, Wu SC, Jordan D, Karvois D, Kamin M. Efficacy and tolerability of topiramate 200 mg/d in the prevention of migraine with/without aura in adults: a randomized, placebo-controlled, double-blind, 12-week pilot study. Clin Ther. 2006 Jul;28(7):1002-11. doi: 10.1016/j.clinthera.2006.07.003. PMID 16990078